CLINICAL TRIAL: NCT01396590
Title: A Randomized, Open-label, Crossover Study to Demonstrate Bioequivalence Between 6 ? 2-mg Tablets of Perampanel and a Single 12-mg Tablet of Perampanel in Healthy Subjects
Brief Title: Demonstrate Bioequivalence Between 6 ? 2-mg Tablets of Perampanel and a Single 12-mg Tablet of Perampanel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2007-A001-040
Record Dates: First submitted 2011-07-13; First posted 2011-07-19 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Central Nervous System
MeSH Terms: interventions — perampanel

ARMS (2):
- 6 x 2 mg perampanel (Active Comparator)
  Interventions: Drug: Perampanel
- 12 mg Perampanel (Active Comparator)
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — 6 x 2 mg perampanel once per day
  Arms: 6 x 2 mg perampanel
Drug: Perampanel — 12 mg perampanel once per day
  Arms: 12 mg Perampanel

SUMMARY:
The purpose of this study is to determine that six 2-mg tablets of perampanel are bioequivalent to one 12-mg tablet of perampanel.

ELIGIBILITY:
Inclusion:

1. Healthy male or female subjects, age 18 to 55 years old, inclusive, at Screening
2. Body mass index (BMI) of 18 to 32 kg/m^2, inclusive, at Screening

Exclusion:

1. Subjects who are taking any prescribed or over-the-counter drug or herbal remedies in the 2 weeks prior to Screening (unless the OTC drug has a long halflife [i.e., 5 x 1/2 greater than 2 weeks]) with the exception of acetaminophen (up to 4 g/day), which is allowed up to 12 hours prior to dosing
2. Subjects who have taken St John's Wort or other dietary aids known to induce CYP3A4 within 4 weeks prior to dosing
3. Subjects who have taken any inhibitor of CYP450 within 2 weeks prior to the first dosing (e.g., grapefruit, grapefruit juice, grapefruit-containing beverages, apple or Seville orange products)
4. Subjects who have received any experimental drug within the 12 weeks leading up to the start of study drug treatment or who are currently enrolled in another clinical trial
5. Subjects with a known or suspected history of alcohol abuse within the 6 months prior to Screening or who have a positive urine drug test or breath alcohol test at Screening or Baseline, or who are unwilling to abstain from consumption of alcohol throughout the periods of in-patient confinement
6. Subjects who consume more than 5 caffeinated beverages per day (e.g., 5 cups of tea, coffee or cans of cola) or who are unwilling to abstain from consumption of caffeine-containing food and beverages throughout the periods of in-patient confinement
7. Subjects who smoke more than 5 cigarettes (or equivalent amount of tobacco) per day or who are unwilling to abstain from the use of nicotine-containing products throughout the period of in-patient confinement
8. Subjects who have a history of drug abuse or dependence or have a positive result from a urine drug screening test
9. Women of child-bearing potential who do not agree to use 2 methods of adequate contraception (e.g., intrauterine device, barrier methods with spermicide) throughout the study and for 30 days after study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cmax of 6 x 2-mg perampanel tablets (reference) compared to that of the 12-mg perampanel tablet (test) | 8 days
AUC(0-t) of 6 x 2-mg perampanel tablets (reference) compared to that of the 12-mg perampanel tablet (test) | 8 days
AUC(0-inf) of 6 x 2-mg perampanel tablets (ref) compared to that of the 12-mg perampanel tablet (test) | 8 days

SECONDARY OUTCOMES:
The incidence of AEs | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cooper, Principal Investigator — Eisai Medical Services
Locations (1):
- Fargo, North Dakota, United States